CLINICAL TRIAL: NCT02111486
Title: A Randomized, Controlled, Cross-over Study of the Effect of Certain Breakfasts on Appetite Control.
Brief Title: Effect of Certain Breakfasts on Appetite Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: St. Boniface Hospital (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Dr. Heather Blewett, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2014:027
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Appetite; Post-prandial Glucose Response
Keywords: Breakfast; Satiety; Fibre; Glucose; Gastric emptying
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- breakfast #1 (Experimental): breakfast food containing high viscosity fibre
  Interventions: Other: breakfast
- breakfast #2 (Experimental): breakfast food containing low viscosity fibre
  Interventions: Other: breakfast
- Control (Placebo Comparator): breakfast food without viscous fibre
  Interventions: Other: breakfast

INTERVENTIONS:
Other: breakfast

SUMMARY:
This clinical trial is being conducted to study whether eating certain meals will reduce your desire to eat and for a longer period of time compared to others and to determine the post-meal glucose response associated with each of these breakfast foods.

DETAILED DESCRIPTION:
The study is divided into 3 phases. Each phase involves eating one of 3 different breakfasts every day for 1 month. The order of the breakfast products is random. During each phase participants will come to the research clinic for 4 visits (1 per week) for assessment of appetite-related sensations. Gastric emptying will be assessed at 1 visit per phase and post prandial glucose response will be measured at 1 visit per phase (Asper site only).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Males and females (not pregnant or lactating) aged 19 to 60 years.
2. Body mass index: 18.5-30 kg/m2.

Exclusion Criteria:

1. A change in medication (dose or type) or medical event requiring hospitalization within the past month.
2. Daily tobacco use.
3. Physical Activity Level >1.8.
4. Eat meals at irregular or unusual times.
5. Food allergy, aversion or unwillingness to eat study foods.
6. Use of any prescription or non-prescription drug, herbal or nutritional supplement known to affect appetite or blood sugar.
7. Presence of a gastrointestinal disorder.
8. Taking drugs that affect gastric emptying.
9. Score >65% on any 1 of the 3 categories of the Three Factor Eating Questionnaire-R18.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Satiety | before the breakfast and every 30 minutes after breakfast for 4 hours
  Total area under the curve (AUC) for hunger, fullness, desire to eat, and prospective consumption scales
Gastric emptying rate | before the breakfast and every 15 minutes after breakfast for 4 hours
  13C-Octanoic Acid will be incorporated into the breakfast food. Rate of gastric emptying will be determined by measuring 13C in breath samples.

SECONDARY OUTCOMES:
Glucose and Insulin | before the breakfast and at 15, 30, 45, 60, 90 and 120 minutes after the the breakfast.
  Total area under the curve (iAUC, mmol*min/L) for both glucose and insulin
Kilocalories | 1 day
  Measure the amount of kilocalories consumed throughout each test day.

OTHER OUTCOMES:
Gastrointestinal side effects | 4 weeks
  Incidence and duration of gastrointestinal side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Blewett, Ph.D, Principal Investigator — I.H. Asper Clinical Research Institute/Agriculture and Agri-Food Canada; Nancy Ames, PhD, Principal Investigator — Richardson Centre for Functional Foods and Nutraceuticals/Agriculture and Agri-Food Canada
Locations (2):
- Canada (2):
  - I.H. Asper Clinical Research Institute, Winnipeg, Manitoba
  - Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba

REFERENCES:
- [Background] Beck EJ, Tosh SM, Batterham MJ, Tapsell LC, Huang XF. Oat beta-glucan increases postprandial cholecystokinin levels, decreases insulin response and extends subjective satiety in overweight subjects. Mol Nutr Food Res. 2009 Oct;53(10):1343-51. doi: 10.1002/mnfr.200800343. PMID 19753601
- [Background] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136
- [Background] Pentikainen S, Karhunen L, Flander L, Katina K, Meynier A, Aymard P, Vinoy S, Poutanen K. Enrichment of biscuits and juice with oat beta-glucan enhances postprandial satiety. Appetite. 2014 Apr;75:150-6. doi: 10.1016/j.appet.2014.01.002. Epub 2014 Jan 14. PMID 24434584
- [Background] Thondre PS, Henry CJ. High-molecular-weight barley beta-glucan in chapatis (unleavened Indian flatbread) lowers glycemic index. Nutr Res. 2009 Jul;29(7):480-6. doi: 10.1016/j.nutres.2009.07.003. PMID 19700035
- [Background] de Graaf C, Blom WA, Smeets PA, Stafleu A, Hendriks HF. Biomarkers of satiation and satiety. Am J Clin Nutr. 2004 Jun;79(6):946-61. doi: 10.1093/ajcn/79.6.946. PMID 15159223